CLINICAL TRIAL: NCT01258699
Title: A Study Comparing the Pharmacokinetics of BK-C-0701 320mg, 480mg and Thiocacid HR Tab 600mg in Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BK-C-0701-101
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-12

CONDITIONS: Healthy Adult Male

ARMS (3):
- 3 (Experimental): BK-C-0701 480mg
  Interventions: Drug: BK-C-0701 480mg
- 2 (Experimental): BK-C-0701 320mg
  Interventions: Drug: BK-C-0701 320mg
- 1 (Active Comparator): Thioctacid HR tab 600mg
  Interventions: Drug: Thiocacid HR Tab 600mg

INTERVENTIONS:
Drug: Thiocacid HR Tab 600mg — 600mg for 1 day
  Arms: 1
Drug: BK-C-0701 320mg — 320mg for 1 day
  Arms: 2
Drug: BK-C-0701 480mg — 480mg for 1 day
  Arms: 3

SUMMARY:
This study is Comparing the Pharmacokinetics of BK-C-0701 320mg, 480mg and Thiocacid HR Tab 600mg in Healthy Adult Male Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male is between 20 and 45
* Weight is between 50 and 90kg, and in 20% of ideal weight. Ideal weight(kg)=(height(cm)-100)*0.9
* Medical history, physical examination, ECG and laboratory test are suitable to the study if judged by an investigator.
* Patient is willing to use an effective method of contraception during the study and for up to 1 months after the use of study drug ceases. (Effective method=spermicide with condom)
* Subject is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

* Patient received drug affected to the study within 14 days from the study initiation.
* Patient received drug-metbolizing enzyme inducer or inhibitor such as Barbiturates within 1 month from the study initiation.
* Subject is hypersensitive investigational drug(Thioctic acid).
* Patient with gastrointestinal history affected absorbing investigational drug or inhibiting normal gastrointestinal motility, gastrointestinal operation or gastrointestinal wound.
* Patient with renal, hepatic, bronchopulmonary, cardiovascular, gastrointestinal, metabolic, neurological, psychotic, oncologic, allergic disease, myocardial infarction, cardiac crisis, hepatitis or pancreatitis history.
* ECG is abnormal.
* Patient abused drug.
* Patient joined other clinical study within 3 months from the study initiation.
* Patient doanted whole blood within 2 months or plasma blood within 1 month from the first medication.
* HBsAg, HCV Ab or HIV Ab are positive.
* Patient who was not suitable to the study if judged by an investigator.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-08

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea